CLINICAL TRIAL: NCT04273373
Title: A Randomized Non-inferiority Trial Comparing Low Dose Albumin Versus Standard Dose Albumin in High Risk Spontaneous Bacterial Peritonitis.
Brief Title: Low Dose Albumin Versus Standard Dose Albumin in High Risk Spontaneous Bacterial Peritonitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-AKI-03
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dose albumin+SOC (Active Comparator): 20% albumin1.5 g/kg at diagnosis and 1 g/kg after 48 hours. SOC (Standard of Care)
  Interventions: Biological: Standard dose Albumin
- Low dose albumin+SOC (Experimental): 20% albumin 0.75 g/kg at diagnosis and 0.5 g/kg. after 48 hours SOC (Standard of Care)
  Interventions: Biological: Low Dose Albumin

INTERVENTIONS:
Biological: Low Dose Albumin — 20% albumin 0.75 g/kg at diagnosis and 0.5 g/kg after 48 hours
  Arms: Low dose albumin+SOC
Biological: Standard dose Albumin — 20% albumin1.5 g/kg at diagnosis and 1 g/kg after 48 hours (duration of infusion 6 hours).
  Arms: Standard dose albumin+SOC

SUMMARY:
AIM:- A randomized non-inferiority trial comparing low dose albumin versus standard dose albumin in high risk Spontaneous Bacterial Peritonitis.

Methodology In this non-inferior randomized controlled trial one group will receive Low dose albumin: 20% albumin 0.75 g/kg at diagnosis and 0.5 g/kg after 48 hours and other group will receive Standard dose albumin: 20% albumin1.5 g/kg at diagnosis and 1 g/kg after 48 h (duration of infusion 6 hours).

Study population: Patients of age > 18 years of age with cirrhosis of liver who are admitted in ward/Intensive Care Unit diagnosed with Spontaneous Bacterial Peritonitis.

Study design: Randomized controlled trial Study period: September 2019- September 2020 Sample size: 300 (150 cases in each group) If there is a true difference in favour of the experimental treatment of 5 % then 270 patients are required to be 80% sure that the upper limit of a one sided 95% confidence interval (or equivalently a 90 % two-sided confidence interval) will exclude a difference in favour of the standard group of more than 5 %. And if the investigators consider 10% drop out final sample size is 270+30=300. 150 in each limb. Cases will be randomly allocated in 2 groups by block randomization method with block size taken as 10.

Monitoring and assessment: all the parameters of the objective and also noted any adverse effects.

Adverse Effects: Nausea, Vomiting, Fever with chills, dyspnea Stopping Rule: in the event of any of the adverse effects during therapy.

Expected Outcome of the project:

Proportion of patients having new development or progression of Acute Kidney Injury by day 7

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Cirrhosis with SBP (community acquired, health care associated and nosocomial) and baseline serum bilirubin ≥4 mg/dl and/or SCr ≥ 1 mg/dl.

Exclusion Criteria:

1. Antibiotic treatment within one week before the diagnosis of SBP (except for prophylactic treatment with norfloxacin)
2. Significant cardiac failure, pulmonary disease
3. Known CKD ( Chronic Kidney Disease)or findings suggestive of organic nephropathy (proteinuria, haematuria, or Abnormal findings on renal USG)
4. Hepatocellular carcinoma
5. HIV (Human Immunodeficiency Virus) infection;
6. GI (Gastrointestinal) bleed within 1 month before the study
7. Ileus
8. Grade 3 to 4 hepatic encephalopathy
9. Other types of infection
10. Shock
11. Presence of any potential causes of dehydration (such as diarrhoea or an intense response to diuretic treatment) within one week before the diagnosis of SBP).
12. Baseline serum bilirubin <4 mg/dl or S. Cr < 1 mg/dl
13. Serum creatinine level of > 3.0 mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having new development or progression of Acute Kidney Injury in both groups | Day 7

SECONDARY OUTCOMES:
Number of participants with resolution of Spontaneous Bacterial Peritonitis in both groups | Day 7
Changes in RRI (Renal Resistive Index) in both groups | Day 6
Number of participants who will develop volume overload in both groups | Day 7
Number of participants who will not survive in both groups. | Day 7
Number of participants who will not survive in both groups. | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Kar PS, Venishetty S, Laroia ST, Jindal A, Maiwall R, Sood AK, Shasthry SM, Rajan V, Arora V, Bhardwaj A, Kumar G, Kumar M. Tolerance of standard dose albumin infused over 6 hrs for treatment of spontaneous bacterial peritonitis-A randomized controlled trial. Indian J Gastroenterol. 2023 Aug;42(4):505-516. doi: 10.1007/s12664-023-01389-x. Epub 2023 Jul 8. PMID 37422602